CLINICAL TRIAL: NCT00360243
Title: 6-mo. Min Eff Dose of Flibanserin: 25 v 50 mg Bid v 50 mg hs v Pbo in Younger Women in NA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sprout Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 511.70
Record Dates: First submitted 2006-08-03; First posted 2006-08-04 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Sexual Dysfunctions, Psychological
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — flibanserin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- flibanserin 25 mg b.i.d (Experimental): 25 mg twice daily for 24 weeks
  Interventions: Drug: flibanserin
- flibanserin 50mg qhs (Experimental): 50 mg taken once daily at bedtime for 24 weeks
  Interventions: Drug: flibanserin
- flibanserin 50mg b.i.d. (Experimental): 50 mg twice daily for 24 weeks
  Interventions: Drug: flibanserin
- placebo (Placebo Comparator): twice daily for 24 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: flibanserin — Experimental: flibanserin 25 mg b.i.d
  Arms: flibanserin 25 mg b.i.d
Drug: flibanserin — Experimental: flibanserin 50mg qhs
  Arms: flibanserin 50mg qhs
Drug: flibanserin — Experimental: flibanserin 50mg b.i.d.
  Arms: flibanserin 50mg b.i.d.
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
This trial is designed to assess the safety and efficacy of flibanserin in the treatment of premenopausal women with Hypoactive Sexual Desire Disorder (HSDD) that meet standard diagnostic criteria. Efficacy for flibanserin will be assessed vs. a parallel placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are 18 years of age and older.
2. Premenopausal women having regular menstrual periods who have HSDD (decreased sexual desire), generalized acquired type, according to DSM IV-TR criteria.
3. Patient must meet minimum cut-off scores on questionnaires relating to sexual functioning and sexual distress.
4. Patients must be willing to try to have sexual activity (e.g., any act involving direct genital stimulation) at least once monthly.
5. Patients must be willing and able to use an electronic diary on a daily basis (e.g., have access to a working land line telephone for daily data transmissions).
6. At the Baseline Visit, patients must have complied with eDiary use adequately.
7. Patients must be in a stable, monogamous, heterosexual relationship that is secure and communicative, for at least 1 year prior to the Screen Visit. The partner is expected to be physically present at least 50% of each month.
8. Patients must have used a medically acceptable method of contraception for at least 3 months before the Baseline Visit (Visit 2) and continue to use that medically acceptable method of contraception during the trial.
9. In the investigators opinion, patients must be reliable, honest, compliant, and agree to co-operate with all trial evaluations as well as to be able to perform them.
10. Patients must be able and willing to give meaningful, written informed consent prior to participation in the trial, in accordance with regulatory requirements. Patients must have sufficient understanding to communicate effectively with the investigator, and be willing to discuss their sexual functioning with the investigative staff.
11. Patients must have a clinically acceptable Pap smear as read by a cytology facility (no evidence of malignancy or squamous intraepithelial lesions) within 6 months before the Screen Visit.

Exclusion Criteria:

1. Patients who have taken any medication noted in the protocols List of Prohibited Medications within 30 days before screening.
2. Patients whose sexual function was affected (enhanced or worsened) in the investigators opinion by any medication within 30 days before the Screen Visit and anytime prior to the Baseline Visit.
3. Patients with a history of drug dependence or abuse within the past one year.
4. Patients with a history of multiple severe reactions (i.e., allergic or oversensitivity to usual doses) to drugs that affect the brain.
5. Patients with a history of participation in a trial of another investigational medication within one month prior to the Screen Visit, or participation in any previous clinical trial of flibanserin.
6. Patients who meet accepted diagnostic criteria for sexual disorders that would interfere with improvement in HSDD (sexual aversion, substance-induced sexual problems, urge to live as a man, etc.
7. Patients who indicate that their sexual partner has inadequately treated sexual problems that could interfere with the patients response to treatment.
8. Patients who have entered the menopausal transition or menopause or have had a hysterectomy.
9. Patients with findings at the Screen Visit of infection, inflammation, undue tenderness, or shrinkage (atrophy) of the female organs.
10. Patients who are breast feeding or have breastfed within the last 6 months prior to the Baseline Visit.
11. Patients who are pregnant or have been pregnant within the last 6 months prior to the Baseline Visit.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1385 (Actual)
Dates: Start 2006-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (81):
- United States (81):
  - 511.70.01068 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 511.70.01040 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 511.70.01041 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 511.70.01003 Boehringer Ingelheim Investigational Site, Jonesboro, Arkansas
  - 511.70.01070 Boehringer Ingelheim Investigational Site, Carmichael, California
  - 511.70.01026 Boehringer Ingelheim Investigational Site, Redding, California
  - 511.70.01015 Boehringer Ingelheim Investigational Site, San Diego, California
  - 511.70.01014 Boehringer Ingelheim Investigational Site, Stanford, California
  - 511.70.01017 Boehringer Ingelheim Investigational Site, Tarzana, California
  - 511.70.01072 Boehringer Ingelheim Investigational Site, Torrance, California
  - 511.70.01078 Boehringer Ingelheim Investigational Site, Vista, California
  - 511.70.01066 Boehringer Ingelheim Investigational Site, Walnut Creek, California
  - 511.70.01064 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 511.70.01001 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 511.70.01050 Boehringer Ingelheim Investigational Site, Farmington, Connecticut
  - 511.70.01006 Boehringer Ingelheim Investigational Site, Hartford, Connecticut
  - 511.70.01055 Boehringer Ingelheim Investigational Site, New London, Connecticut
  - 511.70.01024 Boehringer Ingelheim Investigational Site, Aventura, Florida
  - 511.70.01056 Boehringer Ingelheim Investigational Site, Daytona Beach, Florida
  - 511.70.01090 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 511.70.01027 Boehringer Ingelheim Investigational Site, Gainesville, Florida
  - 511.70.01062 Boehringer Ingelheim Investigational Site, New Port Richey, Florida
  - 511.70.01043 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 511.70.01084 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 511.70.01048 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 511.70.01042 Boehringer Ingelheim Investigational Site, Stuart, Florida
  - 511.70.01063 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 511.70.01085 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 511.70.01086 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 511.70.01022 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 511.70.01057 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 511.70.01087 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 511.70.01052 Boehringer Ingelheim Investigational Site, Roswell, Georgia
  - 511.70.01060 Boehringer Ingelheim Investigational Site, Champaign, Illinois
  - 511.70.01058 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 511.70.01032 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 511.70.01018 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 511.70.01007 Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - 511.70.01047 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 511.70.01079 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 511.70.01031 Boehringer Ingelheim Investigational Site, Saint Louis, Maryland
  - 511.70.01011 Boehringer Ingelheim Investigational Site, Haverhill, Massachusetts
  - 511.70.01028 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 511.70.01081 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 511.70.01082 Boehringer Ingelheim Investigational Site, Billings, Montana
  - 511.70.01077 Boehringer Ingelheim Investigational Site, Moorestown, New Jersey
  - 511.70.01019 Boehringer Ingelheim Investigational Site, Endwell, New York
  - 511.70.01076 Boehringer Ingelheim Investigational Site, New York, New York
  - 511.70.01025 Boehringer Ingelheim Investigational Site, Poughkeepsie, New York
  - 511.70.01067 Boehringer Ingelheim Investigational Site, Purchase, New York
  - 511.70.01016 Boehringer Ingelheim Investigational Site, Mount Airy, North Carolina
  - 511.70.01044 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 511.70.01049 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 511.70.01089 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 511.70.01054 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 511.70.01075 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 511.70.01002 Boehringer Ingelheim Investigational Site, Mayfield Heights, Ohio
  - 511.70.01065 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 511.70.01083 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 511.70.01036 Boehringer Ingelheim Investigational Site, Medford, Oregon
  - 511.70.01004 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 511.70.01021 Boehringer Ingelheim Investigational Site, West Reading, Pennsylvania
  - 511.70.01073 Boehringer Ingelheim Investigational Site, Warwick, Rhode Island
  - 511.70.01023 Boehringer Ingelheim Investigational Site, Anderson, South Carolina
  - 511.70.01035 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 511.70.01008 Boehringer Ingelheim Investigational Site, Nasville, Tennessee
  - 511.70.01020 Boehringer Ingelheim Investigational Site, Corpus Christi, Texas
  - 511.70.01009 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 511.70.01030 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 511.70.01091 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 511.70.01013 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 511.70.01005 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 511.70.01061 Boehringer Ingelheim Investigational Site, Sandy City, Utah
  - 511.70.01010 Boehringer Ingelheim Investigational Site, Burlington, Vermont
  - 511.70.01012 Boehringer Ingelheim Investigational Site, Charlottesville, Virginia
  - 511.70.01046 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 511.70.01029 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 511.70.01071 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 511.70.01033 Boehringer Ingelheim Investigational Site, Bellevue, Washington
  - 511.70.01039 Boehringer Ingelheim Investigational Site, Tacoma, Washington
  - 511.70.01069 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flibanserin 25 mg b.i.d | Flibanserin 50mg Qhs | Flibanserin 50mg b.i.d. | Placebo
Started | 337 | 363 | 336 | 349
Completed | 235 | 243 | 180 | 224
Not Completed | 102 | 120 | 156 | 125

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flibanserin 25 mg b.i.d | Flibanserin 50mg Qhs | Flibanserin 50mg b.i.d. | Placebo | Total
Number analyzed (Participants) | 337 | 363 | 336 | 349 | 1385
Age, Customized [Number; unit: participants]
  18-34 years | 154 | 169 | 145 | 158 | 626
  35-44 years | 153 | 157 | 161 | 164 | 635
  45 years and older | 30 | 37 | 30 | 27 | 124
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 337 | 363 | 336 | 349 | 1385
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White Non Hispanic | 266 | 306 | 276 | 278 | 1126
  White Hispanic | 20 | 20 | 23 | 19 | 82
  Black Non Hispanic | 43 | 31 | 28 | 47 | 149
  Black Hispanic | 2 | 0 | 1 | 2 | 5
  Asian Non Hispanic | 6 | 6 | 7 | 3 | 22
  Asian Hispanic | 0 | 0 | 0 | 0 | 0
  Missing | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to 24 Weeks in the Frequency of Satisfying Sexual Events as Measured by the eDiary.
Description: A small personal handheld electronic device (eDiary) was used by the patients to record information about sexual events. Patients were instructed to complete the eDiary every morning. When completing an eDiary entry, patients answered questions regarding their sexual events since their last eDiary entry. If patients missed or were late with their eDiary entry, they entered information about their sexual events covering a maximum time period of the past 7 days; however, they did not enter any information beyond the last entry.
Time Frame: 24 weeks
Population: The Full Analysis Set (FAS) consisted of those patients who were randomized to a treatment group, received at least one dose of study medication, and had at least one on-treatment efficacy assessment. The FAS was analyzed for efficacy.
Measure: Mean (Standard Deviation); unit: SSEs per week
Arm/Group | Flibanserin 25 mg b.i.d | Flibanserin 50mg Qhs | Flibanserin 50mg b.i.d. | Placebo
Number analyzed (Participants) | 320 | 334 | 291 | 325
SSEs per week | 1.5 (3.4) | 1.6 (4.2) | 1.6 (3.5) | 1.6 (4.3)

2. Primary Outcome: Change From Baseline to 24 Weeks in Responses to the eDiary Daily Desire Question.
Description: Change from baseline in the electronic diary (eDiary) Sexual Desire Monthly Total Score standardized to a 28-day period (total score range 0-84). Change from baseline is calculated as the difference between the four week baseline period and Week 21 to Week 24. Patients were asked to record information daily in the eDiary throughout the trial. Every time the eDiary was completed, a desire question was asked. If a patient did not complete the diary on a given day, the patient was not asked to enter desire information for more than a 24-hour retrospective period. The desire item read "Indicate your most intense level of sexual desire in the last 24 hours / since your last visit." Potential responses included "no," "low," "moderate," or "strong" and was scored 0-3, with 0 indicating no desire and 3 indicating the highest level of desire:
  0 = No desire
  1. = Low desire
  2. = Moderate desire
  3. = Strong desire
Time Frame: baseline to 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Flibanserin 25 mg b.i.d | Flibanserin 50mg Qhs | Flibanserin 50mg b.i.d. | Placebo
Number analyzed (Participants) | 320 | 334 | 291 | 325
units on a scale | 8.8 (0.9) | 7.0 (0.9) | 7.7 (0.9) | 7.5 (0.9)

ADVERSE EVENTS:
Arm/Group | Flibanserin 25 mg b.i.d | Flibanserin 50mg Qhs | Flibanserin 50mg b.i.d. | Placebo
Serious Adverse Events (participants affected / at risk) | 1/337 | 3/363 | 1/336 | 1/349
Other Adverse Events (participants affected / at risk) | 107/337 | 126/363 | 243/336 | 78/349
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin 25 mg b.i.d (N=337) | Flibanserin 50mg Qhs (N=363) | Flibanserin 50mg b.i.d. (N=336) | Placebo (N=349)
Erythema infectiosum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast Cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin 25 mg b.i.d (N=337) | Flibanserin 50mg Qhs (N=363) | Flibanserin 50mg b.i.d. (N=336) | Placebo (N=349)
Somnolence (Nervous system disorders) | 22 (22) | 17 (17) | 58 (58) | 14 (14)
Nausea (Gastrointestinal disorders) | 21 (21) | 26 (26) | 48 (48) | 11 (11)
Dizziness (Nervous system disorders) | 9 (9) | 23 (23) | 57 (57) | 7 (7)
Headache (Nervous system disorders) | 23 (23) | 22 (22) | 26 (26) | 21 (21)
Fatigue (Nervous system disorders) | 11 (11) | 14 (14) | 41 (41) | 9 (9)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 21 (21) | 24 (24) | 13 (13) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No